CLINICAL TRIAL: NCT04677907
Title: Health Economic and Clinical Comparison of Trabecular Metal Uncemented and Cemented Modular Total Knee Replacements - A Double Blinded Randomised Controlled Trial
Brief Title: TRabecular Metal Economic and Clinical Knee Trial
Acronym: TRECK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Zimmer Biomet (Industry); University of Strathclyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GN13OR267
Record Dates: First submitted 2019-04-04; First posted 2020-12-21 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Total Knee Replacement; Orthopedics
Keywords: Total Knee Replacements; Orthopedics; Orthopedic devices; Arthroplasty; Uncemented
MeSH Terms: interventions — Prostheses and Implants

STUDY DESIGN:
Intervention Model Description: A Double Blinded Randomised Controlled Trial
Who Masked: Participant, Care Provider
Masking Description: all blind except surgeon, who will not take part in study or analysis after surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cemented knee replacement (Active Comparator): total knee replacement with cemented modular knee replacement as per current standard for total knee replacements.
  Interventions: Device: Persona (Zimmer) posterior stabilised cemented Trabecular Metal™ (Tibia and Femur) prosthesis
- Uncemented knee replacement (Experimental): total knee replacement with uncemented modular knee replacement, which is CE certified and accepted in the field.
  Interventions: Device: Persona (Zimmer) posterior stabilised uncemented Trabecular Metal™ (Tibia and Femur) prosthesis

INTERVENTIONS:
Device: Persona (Zimmer) posterior stabilised uncemented Trabecular Metal™ (Tibia and Femur) prosthesis — Persona (Zimmer) posterior stabilised uncemented Trabecular Metal™ (Tibia and Femur) prosthesis vs a Persona (Zimmer) posterior stabilised cemented prosthesis
  Arms: Uncemented knee replacement
Device: Persona (Zimmer) posterior stabilised cemented Trabecular Metal™ (Tibia and Femur) prosthesis — Persona (Zimmer) posterior stabilised uncemented Trabecular Metal™ (Tibia and Femur) prosthesis vs a Persona (Zimmer) posterior stabilised cemented prosthesis
  Arms: Cemented knee replacement

SUMMARY:
To compare the differences, if any, in clinical outcome, patient satisfaction and survivorship between cemented and uncemented Total Knee Replacements (TKR)? To investigate if there are health economic implications of using uncemented TKRs in the NHS?

DETAILED DESCRIPTION:
The investigators propose to undertake a randomised controlled trial comparing Trabecular metal uncemented TKR with cemented TKR. The primary aim will be to determine whether there is a clinically significant difference in outcome between cemented and uncemented knee prosthesis over a 10-year period. The investigators will assess the patient's functional ability using two clinical knee scores the New Knee Society Score (NKSS) and Oxford knee score (OKS). In addition to employing these two standard clinical scores, the investigators will also utilise the Forgotten Joint Score (FJS). The FJS differentiates patients' awareness of the participant's artificial joint which is an important concept in knee arthroplasty. In contrast to hip arthroplasty where the majority of patients are unaware of their joint after surgery, knee arthroplasty patients rarely 'forget' that their joint is artificial. Given the difference in physical properties of trabecular metal and standard implants, the FJS scoring system may highlight potential differences that are important to patients and linked to patient satisfaction. Non-subjective assessment will be performed using Inertial Measuring Units (IMU), which measure the relative position of limbs in space and is a useful measure for clinical movement analysis. Participants will be asked to perform daily task such as walking, standing from a chair and walking up and down stairs, wearing the IMU, before and after surgery. This allows us to see functional improvements after surgery and if there are functional differences between the cemented and uncemented implant.

Clinical evaluation and radiological assessment will be carried out over a 10-year period recording complications and clinical performance of patients and implants.

In addition to carrying out a clinical evaluation of the trabecular metal uncemented knee and cemented knee systems, the investigators will also undertake a health economic assessment of the benefits of using uncemented trabecular metal prostheses.

The most expensive resources in a hospital theatre environment are the surgeon and anaesthetist and maximising their utilisation is essential. The removal of cement mixing and curing time from a TKR offers a potential time saving during the operation. However, the time saved using an uncemented prosthesis during a single operation is unlikely, in isolation, to be sufficient to allow additional clinical activity to be carried out. Nevertheless, by combining multiple uncemented knee replacement operations in a single theatre session it may be possible to save sufficient time during the entire day to facilitate an additional surgical procedure, thus increasing the utilisation of surgeons, anaesthetists and theatre staff. If this were achievable, it would add significant value for health care providers.

Despite the success of knee arthroplasty 18% of patients are dissatisfied with their outcome [16]. These are an important group of patients and understanding better the issues that these patients encounter is key in achieving better satisfaction rates and ensuring appropriate use of Orthopaedic implants. The investigators will therefore also study patient factors such as depression and ability to deal with pain/discomfort and correlate these with post-surgical outcome.

Trabecular metal uncemented implants potentially offer benefits to both patient and surgeon but as yet there is insufficient data available to support widespread use of this product. It is the investigators belief that uncemented knees are underutilised by surgeons because there are a number of areas of concern which have not been adequately addressed in clinical studies. The investigators hope to address these concerns in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects may be recruited to the evaluation.
* Age - there are no restrictions relating to age of the patient.
* Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.
* Subjects who in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigation procedures and are willing to return to the hospital for all the required post-operative follow-ups.
* Subjects with uni-lateral osteoarthritis of the knee or subjects with bi-lateral osteoarthritis of the knee, who have a well functioning and pain free knee replacement in the contralateral knee.
* Subjects who require a TKR for surgical management of osteoarthritis

Exclusion Criteria:

* Patients who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in the study.
* Patients with bi-lateral disease that significantly impacts on their current function and pain.
* Patients who require revision knee arthroplasty surgery.
* Disorders of the feet, ankles, hips or spine causing significant abnormal gait or significant pain.
* Neurological conditions affecting movement.
* Patients with a pathology, which, in the opinion of the Chief Investigator, will adversely affect healing.
* Patients with other disorders which, in the opinion of the Chief Investigator, will/could impair rehabilitation.
* Subjects who in the opinion of the study investigator are unlikely to comply with the study follow-up protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2035-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Oxford Knee Score (Patient reported outcome measure of pain and function) | Baseline, 3 months, 1, 2, 5 and 10 years post-operatively
  Oxford Knee Score is a joint specific 12 question questionnaire related to the pain and function participants believe they are experiencing in their affected knee. A score of 0 indicating high pain and poor function, while a score of 48 is a healthy highly functioning knee joint. Oxford Knee Score will be recorded pre-operatively, at 3 months and 1 year post-operatively. The difference measured at 1 year will be the primary outcome. The questionnaire will be completed either, face-to-face, via postal questionnaires or via virtual appointments.

SECONDARY OUTCOMES:
Change in costs per quality adjusted life year (QALY) per participant. | 1, 2 and 10 years post-operatively
  Measured using a breadth of health economic data collected during the course of the study, including, cost of surgery, surgical time, implant costs, other related surgical costs (consumables etc), recovery time, rehabilitation costs, readmissions, revisions surgeries and GP visits in conjunction with quality of life data. This will provide a cost per quality of adjusted life year per participant.
Change in operation time (minutes) | After last intervention is administered
  Measured using video recordings for surgical procedures. Data will be collected from recordings to conduct motion and time analysis to provide an accurate operation time.
Change in clinical movement: walking | Baseline, 3 months, 1, 2 years post-operatively
  Participants will be given an inertial measurement unit which is an electronic device that records movement during an activity.
Change in clinical movement: standing from sitting | Baseline, 3 months, 1, 2 years post-operatively
  Participants will be given an inertial measurement unit which is an electronic device that records movement during an activity.
Change in clinical movement: walking down stairs | Baseline, 3 months, 1, 2 years post-operatively
  Participants will be given an inertial measurement unit which is an electronic device that records movement during an activity.
Change in New Knee Society Score (Patient reported outcome measure of pain and function) | Baseline, 3 months, 1, 2 years' post-operatively
  New Knee Society Score is a validated questionnaire related to the knee pain and function. The questionnaire will be completed either, face-to-face, via postal questionnaires or via virtual appointments.
Change in Forgotten Joint Score (Patient reported outcome measure of their awareness of their artificial knee) | 3 months, 1, 2, 5 and 10 years post-operatively
  Forgotten Joint Score is a validated questionnaire related to the awareness a patients experiences regarding their artificial joint. The questionnaire will be completed either, face-to-face, via postal questionnaires or via virtual appointments.
Change in Patient Satisfaction (Patient reported outcome measure of post-operative satisfaction of the intervention) | 3 months, 1, 2, 5 and 10 years post-operatively
  Patient satisfaction will be reported using a questionnaire asking "Overall, how satisfied are you with the outcome of your surgery?" on a scale of "Very satisfied, satisfied, unsure, dissatisfied and very dissatisfied", and reporting "If you could go back in time, would still chose to have this operation?" as either "Yes or No".
Change in Hospital Anxiety and Depression Score (Patient reported outcome measure of depression and anxiety surrounding hospitalisation) | Baseline, and 1, 2 years' post-operatively
  Hospital Anxiety and Depression Score is a validated 14 point questionnaire related to the a patients anxiety (7 questions) or depression (7 questions) related to hospitalisation. The questionnaire will be completed either, face-to-face, via postal questionnaires or via virtual appointments.
Change in Short Form-12 (Patient reported outcome measure of general quality of life) | Baseline and 1, 2 years post-operatively
  Short form-12 is a validated questionnaire that measures a participants general quality of life. The questionnaire will be completed either, face-to-face, via postal questionnaires or via virtual appointments.
Change in Pain Catastrophising Scale (Patient reported outcome measure of patients perceptions of pain) | Baseline and 1, 2 years' post-operatively
  Pain Catastrophising Scale is a validated questionnaire that reports a patients perception of pain. The questionnaire will be completed either, face-to-face, via postal questionnaires or via virtual appointments.
Change in EuroQoL-5 Dimensions (EQ-5D) (Patient reported outcome measure of a patients perceptions of their overall health) | Baseline, 3 months, 1, 2, 5 and 10 years post-operatively
  EQ-5D is a validated questionnaire that measures an individual's perception of their overall health. The questionnaire will be completed either, face-to-face, via postal questionnaires or via virtual appointments.
Change in Pain Visual Analogue Scale (Patient reported outcome measure of joint pain) | Baseline, 3 months, 1, 2, 5 and 10 years post-operatively
  Pain Visual Analogue Scale is measured on a 100mm scale; 0mm indicating no pain and 100mm indicating worst imaginable pain. The questionnaire will be completed either, face-to-face, via postal questionnaires or via virtual appointments.
Change in Stiffness Visual Analogue Scale (Patient reported outcome measure of joint stiffness) | Baseline, 3 months, 1, 2, 5 and 10 years post-operatively
  Stiffness Visual Analogue Scale is measured on a 100mm scale; 0mm indicating no pain and 100mm indicating worst imaginable pain. The questionnaire will be completed either, face-to-face, via postal questionnaires or via virtual appointments.
Change in Range of Motion (Measure of joint stiffness) | Baseline, 3 months, and 1, 2 years post-operatively
  Range of Motion in the knee is measured using a goniometer. The assessment will be done at a face-to-face appointment by a research nurse.
Change in Post-Op Patient Recovery Diary (Patient Reported outcome measure of pain, stiffness and movement in the immediate post-op period.) | 0 to 6 weeks post-operatively
  Post-Operative Patient Recovery Diaries are completed on daily basis following surgery until 14 days post-operative and subsequently weekly until 6 weeks post-operative. Pain and Stiffness Visual Analogue Scales are measured on a 100mm scale. Patient satisfaction will be reported using a questionnaire asking "Currently how satisfied are you with the pain level of your knee while sitting?" and "Currently how satisfied are you with the pain level of your knee while performing light household duties?" on a scale of "Very Satisfied/Satisfied/Unsure/Dissatisfied/Very dissatisfied". Patient recovery is measured by asking patients "Yes/No" whether they can walked at distance, stand, or walk up and down stairs. In addition, patients are asked for how long they had walked that day before stopping due to pain and on increasing scale of time from 0-5 minutes to >1 hour. Diaries are completed by patients at home.
Change in Canadian Occupational Performance Measure (Patient reported outcome measure of self-perception and performance in everyday living) | Baseline and 1, 2, years' post-operatively
  Canadian Occupational Performance Measure is a validated questionnaire which reports on a participants self-perception and performance in everyday living. The questionnaire will be completed either, face-to-face, via postal questionnaires or via virtual appointments.
Change in PainDETECT Score (Patient reported outcome measure of patients perceptions of pain) | Baseline and 1, 2 years' post-operatively
  PainDETECT Score is a validated questionnaire that reports a patients perception of pain. The questionnaire will be completed either, face-to-face, via postal questionnaires or via virtual appointments.

CONTACTS AND LOCATIONS:
Overall Officials: Mark JG Blyth, Mr, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- Dept of Orthopaedics, Glasgow Royal Infirmary, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen R. A porous tantalum trabecular metal: basic science. Am J Orthop (Belle Mead NJ). 2002 Apr;31(4):216-7. PMID 12008853
- [Background] Hacking SA, Bobyn JD, Toh K, Tanzer M, Krygier JJ. Fibrous tissue ingrowth and attachment to porous tantalum. J Biomed Mater Res. 2000 Dec 15;52(4):631-8. doi: 10.1002/1097-4636(20001215)52:43.0.co;2-6. PMID 11033545
- [Background] Bobyn JD, Stackpool GJ, Hacking SA, Tanzer M, Krygier JJ. Characteristics of bone ingrowth and interface mechanics of a new porous tantalum biomaterial. J Bone Joint Surg Br. 1999 Sep;81(5):907-14. doi: 10.1302/0301-620x.81b5.9283. PMID 10530861
- [Background] Bobyn JD, Toh KK, Hacking SA, Tanzer M, Krygier JJ. Tissue response to porous tantalum acetabular cups: a canine model. J Arthroplasty. 1999 Apr;14(3):347-54. doi: 10.1016/s0883-5403(99)90062-1. PMID 10220190
- [Background] Zardiackas LD, Parsell DE, Dillon LD, Mitchell DW, Nunnery LA, Poggie R. Structure, metallurgy, and mechanical properties of a porous tantalum foam. J Biomed Mater Res. 2001;58(2):180-7. doi: 10.1002/1097-4636(2001)58:23.0.co;2-5. PMID 11241337
- [Background] Gandhi R, Tsvetkov D, Davey JR, Mahomed NN. Survival and clinical function of cemented and uncemented prostheses in total knee replacement: a meta-analysis. J Bone Joint Surg Br. 2009 Jul;91(7):889-95. doi: 10.1302/0301-620X.91B7.21702. PMID 19567852
- [Background] Henricson A, Linder L, Nilsson KG. A trabecular metal tibial component in total knee replacement in patients younger than 60 years: a two-year radiostereophotogrammetric analysis. J Bone Joint Surg Br. 2008 Dec;90(12):1585-93. doi: 10.1302/0301-620X.90B12.20797. PMID 19043129
- [Background] European Training Program in Microseparation Techniques. Methods. 1998 Feb;14(2):235. PMID 9571079
- [Background] Nilsson KG, Karrholm J, Ekelund L, Magnusson P. Evaluation of micromotion in cemented vs uncemented knee arthroplasty in osteoarthrosis and rheumatoid arthritis. Randomized study using roentgen stereophotogrammetric analysis. J Arthroplasty. 1991 Sep;6(3):265-78. doi: 10.1016/s0883-5403(06)80174-9. PMID 1940933
- [Background] Baker PN, van der Meulen JH, Lewsey J, Gregg PJ; National Joint Registry for England and Wales. The role of pain and function in determining patient satisfaction after total knee replacement. Data from the National Joint Registry for England and Wales. J Bone Joint Surg Br. 2007 Jul;89(7):893-900. doi: 10.1302/0301-620X.89B7.19091. PMID 17673581
- See also: Scottish Arthroplasty Report 2018 — https://www.arthro.scot.nhs.uk/docs/2018/2018-08-14-SAP-Annual-Report.pdf?1
- See also: National Joint Registry for England and Wales Annual Report 2018. — https://www.hqip.org.uk/wp-content/uploads/2018/11/NJR-15th-Annual-Report-2018.pdf
- See also: Hip and knee arthroplasty. Australian National Joint Replacement Registry Annual Report 2018 — https://aoanjrr.sahmri.com/documents/10180/576950/Hip%2C%20Knee%20%26%20Shoulder%20Arthroplasty
- See also: Swedish knee arthroplasty register Annual Report 2018. — http://www.myknee.se/en/
- See also: 2004 Report: Total hip and knee replacements in Canada. Canadian Joint replacement Registry (CJRR). — http://publications.gc.ca/collections/Collection/H115-7-2004E.pdf